CLINICAL TRIAL: NCT02630186
Title: A Phase 1b/2 Study of the Safety and Efficacy of Rociletinib (CO-1686) Administered in Combination With MPDL3280A in Patients With Activating EGFR Mutation-positive (EGFRm) Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Phase 1b/2 Study of Safety and Efficacy of Rociletinib in Combination With MPDL3280A in Patients With Advanced or Metastatic EGFR-mutant NSCLC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study terminated before Phase 1 was completed. This study was reprioritized within the rociletinib development program.
Sponsor: Clovis Oncology, Inc. (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO-1686-032
Record Dates: First submitted 2015-12-02; First posted 2015-12-15 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — rociletinib; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm Rociletinib and MPDL3280A (Experimental): Specific doses of rociletinib, taken continuously BID, will be administered in combination with a fixed dose of MPDL3280A, given intravenously on Day 1 of each 21-day cycle.
  Interventions: Drug: Rociletinib; Drug: MPDL3280A

INTERVENTIONS:
Drug: Rociletinib — A novel, potent, covalent (irreversible) small molecule, tyrosine kinase inhibitor (TKI) administered orally (PO) to patients with EGFRm NSCLC.
  Other Names: CO-1686
Drug: MPDL3280A — A human IgG1 monoclonal antibody administered intravenously (IV)
  Other Names: atezolizumab

SUMMARY:
This clinical research study is being carried out in two parts, Phase 1 and Phase 2. The primary purpose of the Phase 1 portion of the study is to observe the safety of the combination of rociletinib and MPDL3280A in EGFR-mutant NSCLC patients.

The primary purpose of the Phase 2 portion of the study is to evaluate the safety and anti-tumor effects of the combination of rociletinib and MPDL3280A, at the best doses for the combination determined in Phase 1, in patients with EGFR-mutant NSCLC.

DETAILED DESCRIPTION:
This is a Phase 1b/2, open-label, non-randomized, multicenter study evaluating the safety and efficacy of rociletinib administered in combination with MPDL3280A.

Phase 1: This will be the dose finding phase of the study. Patients will be enrolled to available Dosing Cohort. Patients who have progressed after prior first- or second-generation EGFR TKI, regardless of T790M mutation status, will be enrolled.

Phase 2: Patients will be enrolled into 2 groups. Group A will enroll eligible first-line patients who are EGFR TKI treatment-naïve and chemotherapy-naïve. Group B will enroll eligible patients who have progressed after prior first- or second-generation EGFR TKI, regardless of T790M mutation status.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status of 0 or 1
* Adequate hematological and biological function, confirmed by defined laboratory values
* Histologically or cytologically documented metastatic or unresectable, locally advanced or metastatic NSCLC, with one or more activating EGFR mutation (eg, G719X, exon 19 deletion, L858R, L861Q) and absence of exon 20 insertion
* Measurable disease as defined by RECIST v1.1
* Biopsy of tumor tissue for central evaluation, within 60 days prior to the first day of study treatment
* For Phase 1 and Phase 2 Group B, progression after prior 1st or 2nd generation EGFR TKI (eg, erlotinib, gefitinib, afatinib). Previous chemotherapy for NSCLC is allowed.
* For Phase 2 Group A, EGFR TKI treatment-naïve and chemotherapy-naïve

Exclusion Criteria:

* Unresolved toxicities from prior therapy
* Symptomatic, untreated or unstable central nervous system or leptomeningeal metastases
* Previous treatment with rociletinib or MPDL3280A, or other 3rd generation EGFR TKI (eg, AZD-9291, HM61713), or PD 1 axis targeted therapy (eg, anti PD 1 or anti-PD L1)
* Prior treatment with CD137 agonists or other immune checkpoint blockade therapies, including anti-CTLA-4 therapeutic antibodies
* Uncontrolled pleural effusion, pericardial effusion or ascites requiring recurrent drainage procedures
* Uncontrolled hypercalcemia or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab (bisphosphonate use for prevention of skeletal events allowed)
* Known hypersensitivity to any component of the MPDL3280A or rociletinib formulations or history or hypersensitivity to chimeric humanized antibodies or fusion proteins
* History of autoimmune disease
* History of prior allogeneic hematopoietic stem cell transplantation or prior solid organ transplantation
* Treatment with systemic immunosuppressive medications within 2 weeks prior to first day of study treatment (inhaled corticosteroids and mineralocorticoids allowed)
* Live attenuated vaccine within 4 weeks prior to first day of study treatment
* Active tuberculosis, active hepatitis, or positive HIV status
* Class II to IV heart failure as defined by the New York Heart Association functional classification system
* Untreated or uncontrolled cardiovascular disease or other symptomatic cardiac dysfunction
* QTCF > 450 ms, inability to measure QT interval on ECG, personal or family history of long QT syndrome, requirement for medications that have the potential to prolong the QT interval
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computerized tomography (CT) scan (history of radiation pneumonitis in radiation field may be allowed)
* Other malignancies within 5 years prior to enrollment, with the exception of carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer, or ductal carcinoma in situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2017-09-05 (Actual); Study Completion 2017-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Rolfe, MD, Study Director — Clovis Oncology, Inc.
Locations (1):
- University of California at Los Angeles, Santa Monica, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three patients were enrolled at a single center in the United States.
Pre-assignment Details: The Dose Finding Phase included a 7 day Run in Period of rociletinib monotherapy, at the Dosing Cohort-defined dose level, prior to the initiation of combination treatment.
Groups:
- Single Arm Rociletinib and MPDL3280A in Combination: Rociletinib (CO-1686), a novel, potent, covalent (irreversible) small molecule, tyrosine kinase inhibitor (TKI) administered orally (PO) to patients with EGFRm NSCLC in combination with MPDL3280A, a human IgG1 monoclonal antibody administered intravenously (IV).
Period: Overall Study
Arm/Group | Single Arm Rociletinib and MPDL3280A in Combination
Started | 3
Completed | 2
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Rociletinib and MPDL3280A in Combination
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 66 [54 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-emergent Adverse Events, as Assessed by NCI CTCAE v4.03
Description: The safety analyses will be performed using the safety population. Safety data analysis will be conducted on all patients receiving at least one dose of rociletinib or MPDL3280A.
Time Frame: Continuously, up to approximately 18.5 months
Population: All patients enrolled in the study.
Measure: Number; unit: Treatment emergent adverse events
Arm/Group | Single Arm Rociletinib and MPDL3280A in Combination
Number analyzed (Participants) | 3
Treatment emergent adverse events | 31

2. Primary Outcome: Maximum Concentration (Cmax) of Rociletinib and Its Metabolites
Description: Blood sampling for PK analyses of both rociletinib and MPDL3280A will be conducted in all patients treated with rociletinib and MPDL3280A. Cmax will be estimated for rociletinib, using non-compartmental models. Comparisons across dose levels will be made to assess proportionality.
Time Frame: Treatment Day 1 and Day 15
Population: Due to the small number of patients enrolled and small number of PK samples collected as a result of early termination of the study, these analyses were not conducted.
Arm/Group | Single Arm Rociletinib and MPDL3280A in Combination
Number analyzed (Participants) | 0

3. Primary Outcome: Time to Maximum Concentration (Tmax) for Rociletinib and Rociletinib Metabolites
Description: Blood sampling for PK analyses of both rociletinib and MPDL3280A will be conducted in all patients treated with rociletinib and MPDL3280A. Tmax will be estimated for rociletinib, using non-compartmental models. Comparisons across dose levels will be made to assess proportionality.
Time Frame: Treatment Day 1 and Day 15
Population: as for outcome 2
Arm/Group | Single Arm Rociletinib and MPDL3280A in Combination
Number analyzed (Participants) | 0

4. Primary Outcome: Minimum Concentration (Cmin) of Rociletinib and Metabolites
Description: Blood sampling for PK analyses of both rociletinib and MPDL3280A will be conducted in all patients treated with rociletinib and MPDL3280A. Cmin will be estimated for rociletinib, using non-compartmental models. Comparisons across dose levels will be made to assess proportionality.
Time Frame: Approximately every 6 weeks up to 24 months
Population: as for outcome 2
Arm/Group | Single Arm Rociletinib and MPDL3280A in Combination
Number analyzed (Participants) | 0

5. Primary Outcome: Area Under the Curve (AUC) of Rociletinib and Rociletinib Metabolites
Description: Blood sampling for PK analyses of both rociletinib and MPDL3280A will be conducted in all patients treated with rociletinib and MPDL3280A. AUC0 24 will be estimated for rociletinib, using non-compartmental models. Comparisons across dose levels will be made to assess proportionality.
Time Frame: Treatment Day 1 and Day 8
Population: Due to the small number of patients enrolled and small number of PK sample collected as a result of early termination of the study, these analyses were not conducted.
Arm/Group | Single Arm Rociletinib and MPDL3280A in Combination
Number analyzed (Participants) | 0

6. Primary Outcome: Maximum Concentration (Cmax) of MPDL3280A
Description: Blood sampling for PK analyses of both rociletinib and MPDL3280A will be conducted in all patients treated with rociletinib and MPDL3280A. Cmax, for MPDL3280A will be assessed using non-compartmental models. Comparisons across dose levels will be made to assess proportionality.
Time Frame: Cycle 1 Day 1
Population: as for outcome 2
Arm/Group | Single Arm Rociletinib and MPDL3280A in Combination
Number analyzed (Participants) | 0

7. Primary Outcome: Minimum Concentration (Cmin) of MPDL3280A
Description: Blood sampling for PK analyses of both rociletinib and MPDL3280A will be conducted in all patients treated with rociletinib and MPDL3280A. Cmin for MPDL3280A will be assessed using non-compartmental models. Comparisons across dose levels will be made to assess proportionality.
Time Frame: Approximately every 6 weeks up to 24 months
Population: as for outcome 2
Arm/Group | Single Arm Rociletinib and MPDL3280A in Combination
Number analyzed (Participants) | 0

8. Primary Outcome: Objective Response Rate Per RECIST v1.1 in Phase 2
Description: To determine the efficacy of the combination of rociletinib and MPDL3280A based on overall response rate per RECIST v1.1 in the following groups of patients:
  * Group A: Patients with EGFRm advanced or metastatic NSCLC who have not previously received an EGFR TKI or chemotherapy.
  * Group B: Patients with EGFRm advanced or metastatic NSCLC who have progressed on a prior EGFR TKI.
Time Frame: Approximately every 6-9 weeks
Population: Given the early termination of the study and that no patients were enrolled in Phase 2 of the study, no conclusions can be drawn.
Arm/Group | Single Arm Rociletinib and MPDL3280A in Combination
Number analyzed (Participants) | 0

9. Secondary Outcome: Objective Response Rate Per Modified RECIST v1.1, Incorporating Immune-related Criteria, in Phase 2
Description: Conventional response criteria may not be adequate to characterize the antitumor activity of immunotherapeutic agents like MPDL3280A, which can produce delayed responses that may be preceded by initial apparent radiological progression, including the appearance of new lesions. Therefore, modified response criteria have been developed that account for the possible appearance of new lesions and allow radiological progression to be confirmed at a subsequent assessment. In this protocol, patients will be permitted to continue study treatment even after modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria for progressive disease are met if the benefit-risk ratio is judged to be favorable.
  These modified criteria are derived from RECIST version 1.1 (v1.1) conventions and immune related response criteria (irRC).
Time Frame: Approximately every 6-9 weeks, up to 24 months
Population: as for outcome 8
Arm/Group | Single Arm Rociletinib and MPDL3280A in Combination
Number analyzed (Participants) | 0

10. Secondary Outcome: Duration of Response Per RECIST v1.1 and Modified RECIST v1.1, Incorporating Immune-related Criteria, in Phase 2
Description: as for outcome 9
Time Frame: Approximately every 6-9 weeks, up to 24 months
Population: as for outcome 8
Arm/Group | Single Arm Rociletinib and MPDL3280A in Combination
Number analyzed (Participants) | 0

11. Secondary Outcome: Progression-free Survival Per RECIST v1.1 and Modified RECIST v1.1, Incorporating Immune-related Criteria, in Phase 2
Description: as for outcome 9
Time Frame: Approximately every 6-9 weeks, up to 24 months
Population: as for outcome 8
Arm/Group | Single Arm Rociletinib and MPDL3280A in Combination
Number analyzed (Participants) | 0

12. Secondary Outcome: Number of Patients Alive at Study Termination
Description: Patients who received the combination of rociletinib and MPDL3280A alive at the termination of this study.
Time Frame: Up to approximately 18.5 months
Population: Count of the number of enrolled patients alive at study termination.
Measure: Number; unit: participants
Arm/Group | Single Arm Rociletinib and MPDL3280A in Combination
Number analyzed (Participants) | 2
participants | 2

13. Secondary Outcome: Longitudinal Changes in Blood Based Biomarkers (eg, Mutations in EGFR) in ctDNA
Description: Tumor tissue, plasma, and blood specimens will be used for pharmacodynamic assessment of rociletinib and/or MPDL3280A activity, to evaluate the concordance of mutant EGFR detection between tissue and plasma, and to explore biomarkers that may be predictive of response or resistance to rociletinib and/or MPDL3280A. Biomarkers and changes in biomarker status will be investigated for associations with rociletinib and/or MPDL3280A exposure, safety, and clinical activity. Given the limited sample size, no formal statistical analysis is planned.
Time Frame: Blood samples will be collected from each patient approximately every 3 weeks, up to 24 months
Population: Due to the small number of patients enrolled and small number of samples collected as a result of early termination of the study, these analyses were not conducted.
Arm/Group | Single Arm Rociletinib and MPDL3280A in Combination
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the date of first dose of study drug and until 28 days after the last dose of study drug.
Description: One patient withdrew consent during the washout period having only received rociletinib. This patient did not receive MPDL3280A.
Arm/Group | Single Arm Rociletinib and MPDL3280A in Combination
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Rociletinib and MPDL3280A in Combination (N=3)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Rociletinib and MPDL3280A in Combination (N=3)
Nausea (Gastrointestinal disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Increased Blood Sugar (Investigations) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Stomach Pain (Investigations) | 1 (1)
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 2 (2)
Weight decreased (Investigations) | 1 (1)
Prolonged QTc interval (Investigations) | 1 (2)
Cellulitis (Infections and infestations) | 1 (1)
Intermittent epigastric discomfort (Investigations) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Epigastric pain (Gastrointestinal disorders) | 1 (1)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1)
Bilateral hearing loss (Ear and labyrinth disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Dysuria (Renal and urinary disorders) | 1 (1)
Firm raised lesion, dorsum of left foot (Skin and subcutaneous tissue disorders) | 1 (1)
Cataracts (Eye disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Swelling finger (General disorders) | 1 (1)
Elevated aspartate aminotransferase (Investigations) | 1 (1)
Elevated alanine aminotransferase (Investigations) | 1 (1)
Elevated blood alkaline phosphatase (Investigations) | 1 (1)
Herpes virus reactivation (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early which lead to small number of subjects analyzed. The study did not reach the target number of participants needed to achieve target power and statistically reliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-26): https://cdn.clinicaltrials.gov/large-docs/86/NCT02630186/Prot_SAP_000.pdf